CLINICAL TRIAL: NCT05433961
Title: Functional and Structural Assessment of Endobronchial Valve Recipients Using Dynamic Hyperpolarized Xenon-129 MRI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Regulatory Compliance
Sponsor: Xemed LLC (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8511358
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: endobroncial valve; hyperpolarized xenon; lung MRI
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hyperpolarized Xenon MRI assessment of lung function in endobronchial valve treated COPD patients (Experimental): Volunteer patients scheduled for receiving endobronchial valve treatment as part of clinical care will be imaged with hyperpolarized xenon prior and post EBV for assessing lung function and improvement.
  Interventions: Drug: MagniXene Hyperpolarized Xenon MRI

INTERVENTIONS:
Drug: MagniXene Hyperpolarized Xenon MRI — Magnetic Resonance Imaging of lung function using Hyperpolarized Xenon as a contrast agent.

SUMMARY:
This study proposes to use hyperpolarized xenon-129 Magnetic Resonance Imaging (MRI) to study lung function of COPD patients who will receive endobronchial valve (EBV) therapy as part of their clinical standard-of-care. Once inhaled, HP xenon can provide information to imagers regarding functionality across specific regions of the lungs through the assessment of the replacement of air during the normal breathing cycle, how much oxygen is in the airspaces, and if the normal spongy tissue structure has been compromised by lung disease. Pre- (baseline) and post-EBV (follow-up) lung function imaging with HPXe will potentially lead to be better understand disease progression and treatment mechanism.

DETAILED DESCRIPTION:
This study will be assessing the pulmonary function of COPD patients receiving endobronchial valve (EBV) therapy as part of their clinical care by using HP 129Xe MRI in an effort to evaluate the imaging technique's performance in identifying abnormal lung function and micromorphology in patients receiving this therapy. HP Xe MRI study visits will last 1-2 hours for each subject, with the possibility of multiple follow-ups in longitudinal studies. The investigators plan to recruit volunteer patients who are scheduled to receive EBV therapy for the treatment of COPD as part of their clinical standard-of-care. Patients will be imaged at at least two time point, pre-EBV (baseline), and ~45 days post-EBV (follow-up).

Subjects will provide a brief medical history and perform pulmonary function testing (PFT) prior to inhalation of HP xenon-129. If a subject has performed a PFT at the Hospital of the University of Pennsylvania or Temple University Hospital within one month of the study visit and the results are accessible by the research team, subjects will not be required to repeat PFTs for the purpose of imaging.

During a typical HXe MRI session, subjects will first be imaged using standard 1H MRI to generate an anatomical reference image. This will be followed by the inhalation of a small amount (~200 ml) of HP 129Xe from a Tedlar™ bag to perform a frequency calibration, as well as determine the effective flip-angle to be used for the subject. Finally, the subject will sequentially inhale up to 50 breaths of hyperpolarized 129Xe from a gas mixing apparatus designed to oxygenate and dilute the gas, maintaining near normoxic conditions and approximately 10% xenon concentration. During this period, the lungs will be continuously imaged using a 3D sequence and a very low flip-angle (~3 degrees) pulse. The subject will be coached to maintain a reasonably steady breathing cadence of 10-15 breaths per minute, depending on their size and natural breathing rate, but will be otherwise unconstrained with respect to breath timing and volume.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients scheduled to receive endobronchial valve therapy
* Patient is conscious, cooperative and agrees to return for scheduled visits and tests

Exclusion Criteria:

* Patients less than 18 years old
* Patients known to be pregnant - a positive pregnancy test will be used to respectively exclude pregnant patients
* Any known contraindication to MRI examination
* Anyone with an implanted metal device
* Inability to provide informed consent
* A language, communication, cognitive or behavioral impairment that might interfere with fully informed participation in the study.
* History of uncompensated organ failure (i.e. organ failure that is not stabilized through medical intervention), which will be assessed by the PI.
* Homelessness or other unstable living situation
* Active drug or alcohol dependence
* Claustrophobia
* Subjects weighting more than 300 pounds.
* Subjects with chest size larger than the bore of MRI machine from the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Lung function changes from baseline (pre) to follow-up (post) EBV procedure as measured with hyperpolarized xenon MRI. | 90 days
  Endobronchial valve receiving patients will have HPXe MRI sessions for assessing lung function parameters as measured from inhaled hyperpolarized xenon distribution inside the lungs. Fractional ventilation will be obtained based on the signal build up for dynamic breathing of HP 129Xe and room air. TV and FRC will be determined based on the signal build up at inhalation and the gas remaining in the lung at exhalation. τ will be determined by the signal intensity reaching other parts of the lung relative to the signal intensity in the trachea. ADC will be determined using diffusion sensitizing gradients according to standard imaging protocols. Additionally, dissolved phase MR imaging of HP 129Xe will be assessed in order to obtain information regarding microstructural abnormalities that affect gas uptake into the blood. All these parameters are mapped as 3D lung images, and they will be compared between baseline and follow-up session.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Ma, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No